CLINICAL TRIAL: NCT06018974
Title: Effectiveness of Digital Gaming Intervention With Yetitablet for Older Peoples' Functioning and Activity in Long-term Care Environment - Quasi-experimental Study
Brief Title: Digital Gaming Intervention for Older People in Long-term Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49/2021
Record Dates: First submitted 2023-08-09; First posted 2023-08-31 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Depressive Symptoms; Aging; Loneliness; Sedentary Behavior; Social Isolation; Physical Inactivity
Keywords: aging; digital games; long-term care; older people; physical functioning; psychological functioning; social functioning; physical activity
MeSH Terms: conditions — Depression; Sedentary Behavior; Social Isolation; Social Adjustment; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yetitablet group (Experimental): Older adults in the experimental group will participate in a 12-week, 3 times per week, 30-60 minutes per session (recommendation) gaming session with Yetitablet in their home facility. Games will be played in group of 3-5 people with participants taking turns. Gaming sessions are supervised by research assistant or facility personnel.
  Interventions: Device: Yetitablet gaming
- Control group (No Intervention): Participants in control group will continue their normal daily activities in their home facility. No intervention is provided to control group (passive control group).

INTERVENTIONS:
Device: Yetitablet gaming — Playing digital games like bowling, memory games, coordination games ect. with the Yetitablet.
  Arms: Yetitablet group

SUMMARY:
Older people in long-term care (LTC) are often less physically active than their community-dwelling peers. Low physical activity level is associated with more symptoms of anxiety and depression as well as with lower physical performance. This weakens coping with daily activities and increases the care costs. Earlier research have found that playing digital games that require physical activity affects positively functioning of older people. Playing can increase physical activity, improve balance and walking speed, lift the mood and create opportunities for social interaction. The effects of digital gaming, especially on objectively measured physical activity and social functioning, are still unclear.

The aim of this study is to evaluate effectiveness of digital gaming intervention with Yetitablet to physical, psychological and social functioning and activity of older people in long-term care environment.

This study investigates the effectiveness of the Yetitablet in improving the functioning of older people. Yetitablet is an assistive technology device developed for special groups. Yetitablet is a large interactive touchscreen tablet with 55" screen and with Android operating system and it includes numerous applications. Yetitablet has mobile stand on wheels, which allows the screen to be raised and lowered, as well as tilted as needed, all the way to a desk position. Applications can be downloaded to the device from the Google Play Store, and it also has its own game applications, such as darts, table hockey and memory game. These games can be played individually or in group. There is no previous scientific research on the effectiveness of the Yetitablet on the functioning and activity of older people in long-term care settings.

DETAILED DESCRIPTION:
Sample size calculation was completed based on an effect size of 0.3 (power = 0.80; α= 0.05). Assuming a 25% attrition rate, a total of 70 residents will be recruited (35 people in a control group and 35 people in the intervention group). Participants will be recruited from LTC facilities for older people in the region of Oulu in northern Finland. Facilities will be selected by purposeful sampling. Participants will be selected by personnel of the facilities purposefully based on the inclusion criteria.

After being informed about the study all suitable residents willing to participate in this study will undergo baseline functional testing on week 0. Same functional measurements will be conducted after three month intervention period. Baseline physical activity will be measured by activity tracker during one week before intervention and during the intervention (3 months). In addition, approximately 10-15 LTC facility personnel will be recruited for semi-structured group interviews to understand more of the effects of Yetitablet to psychological and social functioning as well as social activity of LTC residents. The interviews will also clarify the staff's experiences of using the Yetitablet and its suitability for the everyday life of the facility.

ELIGIBILITY:
Inclusion Criteria:

* lives in a long-term care facility for older people participating in the study
* has sufficient cognitive ability to understand the purpose of the study
* is able to walk (with or without walking aid) the distance required by physical functioning tests (10m)
* no illness restricting light exercise
* no serious, acute illness
* sufficient cognitive skills to understand game instructions
* sufficient functionality of the upper limbs to use the touch screen

Exclusion Criteria:

* unable to move independently even with walking aid
* severe memory disorder or other acute illness
* unable to understand game instructions, or able to concentrate on playing games for the required time
* too weak vision to play games
* unable to use upper limbs to play
* simultaneously receiving some other treatment that differs from usual treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-03-11 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Timed Up and Go test (TUG) at week 12 | Baseline and week 12
  Change in mean scores on the Timed-up-and-Go test (Completion time in seconds, faster performance indicate better functioning).

SECONDARY OUTCOMES:
Change from baseline in the Revised Index for Social Engagement (RISE) at week 12 | Baseline and week 12
  Change in mean RISE points (range 0-6, higher points indicate more social engagement).
Change from baseline in weekly time spent in light to vigorous physical activity | 13 weeks
  Physical activity (weekly time spent in light to vigorous physical activity) measured with wrist-worn physical activity monitor continuously over the 3-month trial
Change in mood before and after every gaming session | Every gaming session during three month long intervention
  Change in mean face scale scores (range 1-5, higher scores indicate better mood).
Change from baseline in hand grip strength at week 12 | Baseline and week 12
  Change in hand grip strength in both hands measured with dynamometer
Change from baseline in the Short Physical Performance Battery (SPPB) at week 12 | Baseline and week 12
  Change in mean scores on the SPPB test (higher scores indicate better functioning).

CONTACTS AND LOCATIONS:
Overall Officials: Satu Elo, PhD, Study Director — Oulu University of Applied Sciences
Locations (1):
- University of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jantunen H, Wasenius N, Salonen MK, Perala MM, Osmond C, Kautiainen H, Simonen M, Pohjolainen P, Kajantie E, Rantanen T, von Bonsdorff MB, Eriksson JG. Objectively measured physical activity and physical performance in old age. Age Ageing. 2017 Mar 1;46(2):232-237. doi: 10.1093/ageing/afw194. PMID 27810849
- [Background] de Oliveira LDSSCB, Souza EC, Rodrigues RAS, Fett CA, Piva AB. The effects of physical activity on anxiety, depression, and quality of life in elderly people living in the community. Trends Psychiatry Psychother. 2019 Jan-Mar;41(1):36-42. doi: 10.1590/2237-6089-2017-0129. Epub 2019 Feb 4. PMID 30994779
- [Background] van Santen J, Droes RM, Holstege M, Henkemans OB, van Rijn A, de Vries R, van Straten A, Meiland F. Effects of Exergaming in People with Dementia: Results of a Systematic Literature Review. J Alzheimers Dis. 2018;63(2):741-760. doi: 10.3233/JAD-170667. PMID 29689716